CLINICAL TRIAL: NCT04461301
Title: Multimodal Prehabilitation for Major Surgery in Elderly Patients to Lower Complications and to Increase Cost Effectiveness: a Randomised, Prospective, Multicenter, Multidisciplinary Trial (PREHABIL Trial).
Brief Title: Multimodal Prehabilitation for Surgery in the Elderly: a Randomised, Prospective, Multicenter, Multidisciplinary Trial
Acronym: PREHABIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Department of clinical research, Bern (Unknown)
Responsible Party: Principal Investigator, Dominique Engel, Dr.med., Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREHAB2020
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-05

CONDITIONS: Frail Elderly Syndrome; Major Surgery
Keywords: Comprehensive Complication Index

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, multi-centre, multidisciplinary, active controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients that meet the inclusion criteria will be randomised and scheduled for surgery at least 2 weeks after the diagnosis/decision to proceed to surgery. This timeframe allows the implementation of a minimal 2 weeks (up to 4 weeks) multidisciplinary prehabilitation program. Prehabilitation program is composed of 4 elements: exercise training, nutritional intervention, correction of anaemia and smoking cessation. An individual treatment strategy will be proposed to the patient by a multidisciplinary team consisting of surgeon, anesthesiologist, dietitian and physiotherapist.
  Interventions: Procedure: Multimodal Prehabilitation
- Control (No Intervention): Perioperative care of the control group will be based on standardized, multi-element, ERAS recommendations as already implemented in the different participating clinics.

INTERVENTIONS:
Procedure: Multimodal Prehabilitation — A multimodal prehabilitation program (exercise, nutrition, anemia correction and smoking cessation).
  Arms: Intervention

SUMMARY:
This multicentric, randomised controlled trial is to the investigators knowledge the first implementation of a multimodal, multidisciplinary prehabilitation approach using knowledge from different specialties to lower complications and to increase cost effectiveness after major surgery in elderly, frail patients.

DETAILED DESCRIPTION:
Postoperative complications occur in up to 50% of patients and major surgery is associated with a 20 to 40% reduction in physiological and functional capacity. The elderly have surgery 4 times more often than the rest of the population, thus in the future a major proportion of patients presenting for surgery will be older than 65 years. Elderly patients have more postoperative complications, a longer convalescence and higher surgical morbidity and mortality. The number and severity of complications are closely related to preoperative functional capacity, nutritional state, psychological state, and smoking behavior. Another population most probably to benefit from such a program are cancer patients with decreased functional health after cancer treatment. Cancer prehabilitation affords an opportunity for the patient to improve functional status while waiting to begin treatment. This is a patient group expected to grow in the future.

This is a multicenter, multidisciplinary, 2 arms (standard, n=233 vs intervention i.e. prehabilitation, n=233), randomised controlled trial (RCT).

The prehabilitation program is composed of 4 elements: exercise training, nutritional intervention, correction of anaemia and smoking cessation.

This multicentric, randomised controlled trial is to the investigators knowledge the first implementation of a multimodal, multidisciplinary prehabilitation approach using knowledge from different specialties to lower complications and to increase cost effectiveness after major surgery in elderly, morbid patients.

The primary outcome is measured by the comprehensive complication index (CCI). Secondary outcomes are physical parameters measured by cardio-pulmonary exercise testing (CPET), grip strengh, Nutritional Risk Score (NRS). Further outcomes are amongst others smoking behavior, haemoglobin concentration, days at home at 30 days (DAH30) and quality of recovery 15 (QoR15).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* comorbid (≥ASA 3)
* pre-existing fitness deficit: AT<11ml/kg/min respectively VO2peak<14ml/kg/min if AT unavailable or VE/VCO2 slope > 33
* scheduled for major urologic, thoracic, visceral, orthopaedic or cardiovascular surgery
* screening at least 2 weeks prior to surgery

Exclusion Criteria:

* Paralysis or patients with mobility problems (who are unable to exercise),
* Premorbid conditions or orthopaedic impairments that contraindicate exercise,
* Cognitive disabilities,
* Chronic renal failure (need for dialysis)
* Emergency procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) | 30 days after surgery
  The comprehensive complication index (value from 0 = no complication to 100 = death) is a valuable, validated index for the assessment of multiple postoperative complications. It has been developed based on Swiss hospital data and has been validated internationally.

SECONDARY OUTCOMES:
Cardiovascular & Pulmonary | Before and after 2-4 weeks of prehabilitation, at 30 days
  Cardio-Pulmonary Exercise Test (CPET): Peak VO2, VO2 at VT1, peak VE, VE/VCO2 slope, O pulse, FEV1, FEV1/FVC, resting HR, HR reserve, resting systolic and diastolic BP, CPAx ICUD and CPAX HosD in case of ICU admission, Maximum inspiratory pressure , Grip strength, NTproBNP, serial hsTroponin in case of raised NTproBNP, change in preoperative P-POSSUM score
Nutrition & Bioimpendance | At the beginning of study, before and after surgery, at 30 days.
  Nutritional Risk Score (NRS), Bio impedance: weight, muscle mass, fat mass, percent body fat, extracellular water/intracellular water, and phase angle, Fat Free Body Mass (FFM) and Lean body Mass (LBM), Days nil per mouth
Anaemia | 30 days after surgery
  Presence of anaemia, Transfusion rates in the first 30 days after surgery.
Smoking | At the beginning of study, before and after surgery, at 30 days.
  Successful smoking cessation rate, Exhaled CO measured.
Questionnaires for recovery, anxiety and cardiac risk | At the beginning of study, before and after surgery, at 30 days.
  Quality of Recovery Score (QoR-15), State-Trait Anxiety Inventory Test (STAI-T), Duke Activity Status Index (DASI)

OTHER OUTCOMES:
Other outcomes of interest | At 30/90 days
  Length of hospital stay, Days at home at 30 days, Predicted costs for visceral interventions, CCI at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dominique A Engel, Dr, Principal Investigator — Department of Anaesthesiology and Pain Therapy, University Hospital Bern
Locations (1):
- Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetsch T, Dueblin SW, Eser P, Beilstein CM, Wuethrich PY, Wilhelm M, Engel D. Effect of multimodal home-based prehabilitation on objectively measured physical activity in patients undergoing elective cardiac or non-cardiac major surgery: secondary outcomes from a randomised controlled trial. Perioper Med (Lond). 2025 Jul 4;14(1):69. doi: 10.1186/s13741-025-00554-4. PMID 40615882
- [Derived] Beilstein CM, Krutkyte G, Vetsch T, Eser P, Wilhelm M, Stanga Z, Bally L, Verra M, Huber M, Wuethrich PY, Engel D. Multimodal prehabilitation for major surgery in elderly patients to lower complications: protocol of a randomised, prospective, multicentre, multidisciplinary trial (PREHABIL Trial). BMJ Open. 2023 Jan 3;13(1):e070253. doi: 10.1136/bmjopen-2022-070253. PMID 36596634